CLINICAL TRIAL: NCT02197234
Title: A Phase I, Open-Label, Non-Randomised, Multicentre Study to Assess the Effect of AZD9291 on the Pharmacokinetics of Simvastatin (a Sensitive CYP3A4 Substrate) in Patients With EGFRm Positive NSCLC Whose Disease Has Progressed on an EGFR TKI
Brief Title: Study to Assess the Effect of AZD9291 on the Blood Levels of Simvastatin in Patients With EGFRm+ NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00014; 2014-002070-36 (EudraCT Number)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: oncology, cancer, non small cell lung cancer, anticancer drug, pharmacokinetics, AZD9291, simvastatin, EGFR genes
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9291 and simvastatin (Experimental): Sequential treatments of simvastatin alone followed by AZD9291 alone, followed by simvastatin + AZD9291.
  Interventions: Procedure: Pharmacokinetic sampling - AZD9291; Drug: Simvastatin; Drug: AZD9291 tablet dosing; Procedure: Pharmacokinetic sampling - simvastatin; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550

INTERVENTIONS:
Procedure: Pharmacokinetic sampling - AZD9291 — Blood sampling to measure AZD9291
Drug: Simvastatin — Simvastatin (CYP substrate) 40mg taken once daily on Days 1 and 31 (Part A)
Drug: AZD9291 tablet dosing — AZD9291 80mg tablet taken from Days 3 to 32. (Part B) AZD9291 80mg tablet taken daily for 12 months.
Procedure: Pharmacokinetic sampling - simvastatin — Blood sampling to measure simvastatin levels
Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550 — Blood samples to measure levels of AZ5140 and AZ7550

SUMMARY:
This is a Phase I, open-label, 2-part study in patients with a confirmed diagnosis of epidermal growth factor receptor (EGFR) mutation positive (EGFRm+) non-small cell lung cancer (NSCLC), who have progressed following prior therapy with an approved EGFR tyrosine kinase inhibitor (TKI) agent.

Part A will assess the effect of AZD9291 on the pharmacokinetic (PK) parameters of simvastatin and simvastatin acid, following multiple oral dosing of AZD9291 in a fasted state.

Part B will allow patients further access to AZD9291 after the PK phase (Part A) and will provide for additional safety data collection. All patients from Part A who completed treatment may continue to receive AZD9291 80 mg once daily until: disease progression; they are no longer deriving clinical benefit; or any other reason.

ELIGIBILITY:
For inclusion in the study patient should fulfil the following criteria:

1. Male or female, aged at least 18 years.
2. Histological or cytological confirmation diagnosis of NSCLC.
3. Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI, eg gefitinib, afatinib or erlotinib. In addition, other lines of therapy may have been given. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study.
4. Confirmation that the tumour harbours an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 with no deterioration over the previous 2 weeks (Appendix G).
6. Patients must have a life expectancy of ≥12 weeks as estimated at the time of screening.
7. Females should be using adequate contraceptive measures and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments; women under 50 years old would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution; documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.
8. Male patients should be willing to use barrier contraception, ie, condoms, until 6 months after last study drug is taken.

Exclusion criteria:

1. Participation in another study with an IP during the last 14 days (or a longer period depending on the defined characteristics of the agents used).
2. Treatment with any of the following: Treatment with an EGFR TKI (eg, erlotinib or gefitinib) within 8 days or approx. 5 x half-life, whichever is the longer, of the first dose of study treatment; any cytotoxic chemotherapy, investigational agents or other anticancer drugs from a previous treatment regimen or clinical study within 14 days of the first dose; major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment; radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose; patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inhibitors of CYP3A4 (at least 1 week prior) and potent inducers of CYP3A4 (at least 3 week prior). All patients must avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4.
3. Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
4. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of the IP until the final PK sample collection on Day 32 of Part A.
5. Spinal cord compression or brain metastases unless asymptomatic, stable and not requiring steroids for at least 4 weeks prior to start of study treatment.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the PI's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C, and HIV. Screening for chronic conditions not required.
7. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values: ANC <1.5 x 10^9/L; platelet count <100 x 10^9/L; haemoglobin <90 g/L; ALT >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases; Aspartate aminotransferase (AST) >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases; total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or liver metastases; creatinine >1.5 times ULN concurrent with creatinine clearance <50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
8. Any of the following cardiac criteria: mean resting corrected QT interval corrected for heart rate using Fridericia's correction factor (QTcF) >470 msec obtained from 3 ECGs; any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec; any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under age of 40 or any concomitant medication known to prolong the QT interval.
9. Patients unable to swallow oral medication or patients with GI disorders or significant GI resection likely to interfere with the absorption of AZD9291.
10. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
11. Women who are breastfeeding.
12. Patients with a known hypersensitivity to AZD9291, simvastatin, or any of the excipients of the products.
13. Concomitant medication contraindicated for use with simvastatin due to drug interaction associated with increased risk of rhabdomyolysis (including, but not limited to): itraconazole, ketoconazole, posaconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors (eg, nelfinavir), nefazodone, cyclosporine, danazol, gemfibrozil, amiodarone, amlodipine.
14. 3-hydroxy-3-methyl-glutaryl coenzyme A (HMG-CoA)-reductase inhibitors, such as lovastatin and simvastatin.
15. For optional genetic research: Previous allogenic bone marrow transplant or non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-12-22 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ghiorghiu, MSD, Study Director — AstraZeneca
Locations (13):
- Research Site, Atlanta, Georgia, United States
- Research Site, Leuven, Belgium
- France (5):
  - Research Site, Angers
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Rennes
  - Research Site, Saint-Herblain
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (4):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Harvey RD, Aransay NR, Isambert N, Lee JS, Arkenau T, Vansteenkiste J, Dickinson PA, Bui K, Weilert D, So K, Thomas K, Vishwanathan K. Effect of multiple-dose osimertinib on the pharmacokinetics of simvastatin and rosuvastatin. Br J Clin Pharmacol. 2018 Dec;84(12):2877-2888. doi: 10.1111/bcp.13753. Epub 2018 Oct 10. PMID 30171779
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00014&attachmentIdentifier=29f78d94-42f1-438b-8725-9b62e85740a1&fileName=D5160C00014_study-synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 22 December 2014; Last Subject Last Visit Part A: 30 April 2015 and Part B: 13 May 2016. Study performed at 17 sites across Asia, North America and Western Europe. Part A assessed effect of multiple doses of AZD9291 on PK of simvastatin; Part B allowed subjects further access to AZD9291 and provided additional safety data.
Pre-assignment Details: 57 patients were enrolled (signed informed consent). Patients were assigned to treatment if they met all the inclusion and none of the exclusion criteria. 5 patients were enrolled but failed inclusion/exclusion criteria and so were not eligible to be assigned treatment. The remaining 52 patients started Period 1 and received treatment.
Groups:
- Simvastatin and AZD9291 (Part A); AZD9291 Alone (Part B): In Part A of the study, sequential treatments of simvastatin alone followed by AZD9291 alone, followed by simvastatin + AZD9291. Each patient received 80 mg oral doses of AZD9291 tablets once daily for 30 days (Days 3 to 32) and single 40 mg oral doses of simvastatin on Day 1 and Day 31.
  In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Period: Part A: Day 1-2 (Simvastatin Alone)
Arm/Group | Simvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Started | 52
Completed | 52
Not Completed | 0
Period: Part A: Day 3-30 (AZD9291 Alone)
Arm/Group | Simvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Started | 52
Completed | 50
Not Completed | 2
Not completed — Condition under investigation worsened | 1
Not completed — Withdrawal by Subject | 1
Period: Part A: Day 31-32 (Simvastatin+AZD9291)
Arm/Group | Simvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Started | 49
Completed | 49
Not Completed | 0
Period: Part B: Day 33 to End Part B (AZD9291)
Arm/Group | Simvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Started | 50 (49 completed Part A + 1 entered Part B without completing Part A (due to AE) = 50 started Part B)
Completed | 20
Not Completed | 30
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 6
Not completed — Condition under investigation worsened | 22

BASELINE CHARACTERISTICS:
Arm/Group | Simvastatin and AZD9291 (Part A); AZD9291 Alone (Part B)
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Simvastatin
Description: Pharmacokinetics of simvastatin by assessment of maximum plasma simvastatin concentration
Time Frame: Blood samples collected on Days 1 and 31 at pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 28, and 32 hours post simvastatin dose in Part A
Population: Pharmacokinetic population - all patients who received at least 1 dose of simvastatin or AZD9291 and had at least 1 postdose PK measurement without important protocol deviations/violations.
Measure: Geometric Mean (Full Range); unit: ng/mL
Groups:
- Simvastatin Alone: Simvastatin (CYP substrate) 40mg taken as single dose on Day 1.
- AZD9291 + Simvastatin: AZD9291 80 mg once daily on Days 3 to 32; Simvastatin 40 mg on Day 31.
Arm/Group | Simvastatin Alone | AZD9291 + Simvastatin
Number analyzed (Participants) | 46 | 43
ng/mL | 24.54 [2.69 to 75.5] | 18.65 [3.87 to 141]
Statistical Analysis 1: Comparison: Simvastatin Alone vs AZD9291 + Simvastatin; Study sized so experiment-wise power for the 90% CIs of geometric mean ratios for both AUC and Cmax of AUC9291 being within 70-143% was 90% (95% for each parameter). Within patient CV assumed to be 45%. No change in exposure was also assumed; Test type: Non-Inferiority or Equivalence — 90% CIs being within 70% to 143%; Geometric mean ratio = 77.08, 90% CI 2-sided [63.41 to 93.70] — Simvastatin + AZD9291 / Simvastatin alone. Based on linear mixed-effects model with treatment as fixed effect and patient as a random effect

2. Primary Outcome: AUC of Simvastatin
Description: Pharmacokinetics of simvastatin by assessment of area under the plasma concentration time curve from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng.h/mL
Arm/Group | Simvastatin Alone | AZD9291 + Simvastatin
Number analyzed (Participants) | 46 | 41
ng.h/mL | 80.25 [23.9 to 289] | 73.54 [25.2 to 488]
Statistical Analysis 1: Comparison: Simvastatin Alone vs AZD9291 + Simvastatin; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — 90% CIs being within 70% to 143%; Geometric mean ratio = 91.46, 90% CI 2-sided [77.16 to 108.41] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Tmax of Simvastatin and Simvastatin Acid
Description: Pharmacokinetics of simvastatin and simvastatin acid by time to Cmax
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Simvastatin Alone | AZD9291 + Simvastatin
Number analyzed (Participants) | 46 | 43
hours
  Simvastatin | 1.50 [0.45 to 4.00] | 1.50 [0.50 to 10.00]
  Simvastatin acid | 3.08 [0.50 to 10.00] | 3.08 [1.50 to 12.45]

4. Secondary Outcome: CL/F of Simvastatin
Description: Rate and extent of absorption of simvastatin by assessment of apparent clearance following oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | Simvastatin Alone | AZD9291 + Simvastatin
Number analyzed (Participants) | 46 | 41
L/h | 498.3 [138 to 1670] | 543.9 [82.0 to 1590]

5. Secondary Outcome: Cmax of Simvastatin Acid
Description: Pharmacokinetics of simvastatin acid by assessment of maximum plasma simvastatin acid concentration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Simvastatin Alone | AZD9291 + Simvastatin
Number analyzed (Participants) | 46 | 43
ng/mL | 4.187 [0.482 to 68.5] | 4.161 [0.849 to 66.9]

6. Secondary Outcome: AUC of Simvastatin Acid
Description: Pharmacokinetics of simvastatin acid by assessment of area under the plasma concentration time curve from zero to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng.h/mL
Arm/Group | Simvastatin Alone | AZD9291 + Simvastatin
Number analyzed (Participants) | 42 | 37
ng.h/mL | 31.18 [6.19 to 436] | 30.16 [6.69 to 443]

7. Secondary Outcome: AUC(0-t) of Simvastatin and Simvastatin Acid
Description: Pharmacokinetics of simvastatin and simvastatin acid by assessment of area under the plasma concentration time curve from time zero to last quantifiable dose
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ng.h/mL
Arm/Group | Simvastatin Alone | AZD9291 + Simvastatin
Number analyzed (Participants) | 46 | 43
ng.h/mL
  Simvastatin | 77.97 [21.6 to 279] | 70.17 [24.9 to 470]
  Simvastatin acid | 29.25 [5.71 to 435] | 29.60 [6.34 to 442]

ADVERSE EVENTS:
Time Frame: Approximately 1 month for Part A; up to approximately 14 months for Part B and approximately 15 months for Overall (Parts A and B combined).
Description: Part A: Adverse events (AEs) collected from day of first dose until day prior to first dose in Part B (Day 33), or until 30 days after last dose if discontinued in Part A.
  Part B: AEs collected from day of first dose in Part B until 30 days after last dose, or until last dose in Part B for those entering continued access phase (CAP).
Groups:
- Overall Safety Population: Parts A and B of the study combined.
- Part A Safety Population: In Part A of the study, each patient received 80 mg oral doses of AZD9291 tablets once daily for 30 days (Days 3 to 32) and single 40 mg oral doses of simvastatin on Day 1 and Day 31.
- Part B Safety Population: In Part B of the study, each patient received 80 mg oral AZD9291 tablet formulation once daily, for the duration of their participation.
Arm/Group | Overall Safety Population | Part A Safety Population | Part B Safety Population
All-Cause Mortality (participants affected / at risk) | 5/52 | 0/52 | 8/50
Serious Adverse Events (participants affected / at risk) | 11/52 | 4/52 | 8/50
Other Adverse Events (participants affected / at risk) | 50/52 | 39/52 | 45/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Safety Population (N=52) | Part A Safety Population (N=52) | Part B Safety Population (N=50)
Bundle branch block left (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — Death
Infectious pleural effusion (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) — Death
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Death (same subject as Respiratory failure fatal outcome SAE)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) — Death (same subject as Pneumonia aspiration fatal outcome SAE)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Safety Population (N=52) | Part A Safety Population (N=52) | Part B Safety Population (N=50)
Anaemia (Blood and lymphatic system disorders) | 6 (8) | 2 (2) | 5 (6)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 2 (2) | 3 (5)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 1 (1) | 4 (5)
Constipation (Gastrointestinal disorders) | 9 (12) | 4 (4) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 21 (22) | 8 (9) | 13 (13)
Nausea (Gastrointestinal disorders) | 11 (14) | 6 (6) | 8 (8)
Stomatitis (Gastrointestinal disorders) | 4 (6) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1) | 5 (5)
Asthenia (General disorders) | 11 (22) | 4 (4) | 9 (18)
Fatigue (General disorders) | 10 (11) | 4 (4) | 7 (7)
Non-cardiac chest pain (General disorders) | 4 (5) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 7 (9) | 3 (3) | 4 (6)
Xerosis (General disorders) | 5 (5) | 5 (5) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 7 (7) | 2 (2) | 5 (5)
Paronychia (Infections and infestations) | 11 (16) | 3 (3) | 8 (13)
Respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 3 (4) | 0 (0) | 3 (4)
Blood creatinine increased (Investigations) | 5 (5) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 12 (15) | 5 (5) | 7 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (10) | 1 (1) | 9 (9)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 8 (8) | 2 (2) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (4) | 0 (0) | 3 (4)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3) | 2 (2)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 4 (4) | 14 (17)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (3) | 3 (3)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 3 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 6 (6)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 (12) | 4 (4) | 5 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (19) | 6 (6) | 9 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (4) | 5 (5)
Rash macular (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2) | 4 (4)
Rash papular (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 4 (4) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
At end of Part B, the CAP allowed patients to continue receiving AZD9291 if still deriving clinical benefit. No clinical data was databased during the CAP; thus AE data is presented to end of Part B only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent application.